CLINICAL TRIAL: NCT05244018
Title: Outcome of High Dose Vitamin D on Prognosis of Sepsis Requiring Mechanical Ventilation; A Randomized Controlled Trial
Brief Title: Outcome of High Dose Vitamin D on Prognosis of Sepsis Requiring Mechanical Ventilation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, Assistant Professor of Anesthesia and Intensive Care Department, Faculty of Medicine, Ain- shams University, Cairo, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MS 47/ 2022
Record Dates: First submitted 2022-01-29; First posted 2022-02-17 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1(Treatment group) (Active Comparator)
  Interventions: Drug: Vitamin D3 tablets
- Group 2(Control group) (Active Comparator)
  Interventions: Drug: Vitamin D tablets

INTERVENTIONS:
Drug: Vitamin D3 tablets — Vitamin D3 tablets 50,000 IU units
  Arms: Group 1(Treatment group)
Drug: Vitamin D tablets — Vitamin D tablets 5000 units as daily requirements
  Arms: Group 2(Control group)

SUMMARY:
There is a high prevalence of vitamin D deficiency in the critically ill patient population, with approximately 60% of patients found to be vitamin D deficient, (25(OH)D concentrations <20 ng/mL) and an additional 30% of patients being vitamin D insufficient, (25(OH)D = 20-30 ng/mL).Approximately 80% of sepsis/septic shock patients experience respiratory failure and require mechanical ventilation. Furthermore, several studies document that vitamin D deficiency could be associated with poor outcomes in critically ill patient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with sepsis and required mechanical ventilation (MV) within 24 hours from ICU admission.
* Expected to require mechanical ventilation for at least 72 hours after study entry.

Exclusion Criteria:

* Age <18 years.
* inability to obtain informed consent from the patient and/or legally authorized representative.
* BMI> 40.
* Pregnant or breastfeeding.
* Chronic kidney diseases
* Pancreatitis.
* Hepatic insufficiency
* Cases with coagulopathy
* Moribund and not expected to survive 96 hours.
* Ongoing shock
* History of therapy with high dose vitamin D3 within previous 6 months.
* History of disorders associated with hypercalcemia
* Cancer as the cause of sepsis.
* Subjects undergoing chemotherapy.
* Immune compromised patients.
* Pneumonia developed < 48 hours following intubation.
* Patients with history of aspiration before intubation.
* known allergy to vitamin D.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in procalcitonin level (ng/ml) and antimicrobial peptide cathelicidin (LL37) (ng/ml) level at day 7. | 7 days
  Change in procalcitonin level (ng/ml) and antimicrobial peptide cathelicidin (LL37) (ng/ml) level at day 7.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University Hospitals, Cairo, Egypt